CLINICAL TRIAL: NCT03064880
Title: Does Preoperative Maximization Fluid Strategies for Goal-directed Therapy Affect Physiological Changes Following One-lung Ventilation
Brief Title: Preoperative Goal-directed Fluid Therapy and Physiological Changes Following One-lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201605133RINB
Record Dates: First submitted 2017-02-01; First posted 2017-02-27 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Therapy Adverse Effect
Keywords: Thoracic surgery; Fluid responsiveness; Hemodynamics; Oxidative stress; Goal-directed fluid therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SV maximization (Active Comparator): Dynamic fluid responsiveness parameters, such as stroke volume (SV) response to fluid therapy, are precise fluid indicators that specifically determine patient volume status and are helpful for clinicians to determine the appropriate time for fluid bolus. For SV maximization, the investigators maximize SV after anesthetic induction by fluid therapy up to achieve maximized SV maintained.
  Interventions: Other: SV maximization
- SV normalization (No Intervention): NO active fluid therapy.

INTERVENTIONS:
Other: SV maximization — Voluven solution 250 mL infusion per 5 minutes up to the platau of Flank-starling law: status to SV change < 10% and maintained for 20 minutes
  Arms: SV maximization

SUMMARY:
Intraoperative goal-directed fluid therapy (GDFT) is proposed to improve the outcomes of patients undergoing major surgery. In the GDFT algorithm, the employment of fluid bolus plays a crucial role. Dynamic fluid responsiveness parameters, such as stroke volume (SV) response to fluid infusion, are precise fluid indicators that specifically determine patient volume status and are helpful for clinicians to determine the appropriate time for fluid bolus. In this study, we compared two fluid strategies guided by SV response, namely maximization and nonmaximization protocols, during intraoperative GDFT for patients undergoing thoracic surgery requiring one-lung ventilation. Clinical outcomes and perioperative changes in serum biomarkers of oxidative injury were compared between the two groups as the primary and secondary outcomes respectively.

DETAILED DESCRIPTION:
Intraoperative goal-directed fluid therapy (GDFT) is proposed to improve the outcomes of patients undergoing major surgery. In the GDFT algorithm, the employment of fluid bolus plays a crucial role. Dynamic fluid responsiveness parameters, such as stroke volume (SV) response and stroke volume variation (SVV), are precise fluid indicators that specifically determine patient volume status and are helpful for clinicians to determine the appropriate time for fluid bolus. During GDFT, fluid is commonly administered to maximize perfusion by maintaining patient blood volume at the plateau portion of the Frank-Starling curve by keeping patient at a lower SV response (i.e., SV increase < 10% and maintained for 20 minutes). However, maximization does not necessarily imply optimization; the role of fluid maximization of perfusion in GDFT remains controversial.Moreover, the importance of intraoperative GDFT in thoracic surgery has rarely been explored, because most intraoperative GDFTs have been conducted during abdominal surgery. Acute lung injury (ALI) following thoracic surgery remains a major source of morbidity and mortality after lung resection. Despite the advancement in both the surgical techniques and the perioperative management, the incidence of postoperative ALI remains remarkable. Risk factors are evident, including preoperative pulmonary function, type of surgical procedure, intraoperative fluid management, one-lung ventilation, and ventilator settings. Fluid management for thoracic surgery is challenging. Evidence has shown the association between excessive fluid administration and development of acute lung injury. Therefore, fluid restriction may benefit patients undergoing thoracic surgery. By contrast, restrictive fluid management incurs risks such as a hypovolemic state with impaired tissue perfusion which may result in organ dysfunction and in particular postoperative acute kidney injury. Accordingly, maintenance of perfusion through a maximized fluid protocol may be favorable. However, this debate has not yet been investigated.In this study, two fluid strategies guided by SV response, namely maximization and nonmaximization protocols, during intraoperative GDFT for patients undergoing thoracic surgery requiring one-lung ventilation. Clinical outcomes and perioperative changes in serum biomarkers of oxidative injury were compared between the two groups as the primary and secondary outcomes respectively.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic patients requiring thoracic surgery and lung isolation
* Age 20 - 70 years old

Exclusion Criteria:

* Arrhythmia and irregular heart beats
* End-stage organ disease and difficult to manipulate fluid status
* Pregnant women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-15 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes (postoperative) | 1 year
  collected from chart review including feeding time(hrs postop), hospitalization (days) ICU stay(hrs), any cardiac, pulmonary, and other major organ complications up to 12 months
intraoperative physiological changes and managements | 1day
  collected from anesthetic record including blood pressure changes(mmHg), data from arterial blood gas, use of vasoconstrictors, etc.,

SECONDARY OUTCOMES:
Perioperative oxidative injury biomarkers | 1 day
  tests on intraoperative serum sample, including baseline after anesthetic induction, during one lung ventilation, and resuming two lung ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, MD, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: Undecided